CLINICAL TRIAL: NCT03140852
Title: Community-Based Continence Promotion: Sustaining Healthy Aging in Place (SHAIP) Through Mind Over Matter (MOM)
Acronym: SHAIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0133; A532840 (Other: UW Madison); SMPH\OBSTET & GYNECOL\RESEARCH (Other: UW Madison); 4K12DK100022 (NIH)
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2019-12

CONDITIONS: Fecal Incontinence in Old Age; Urinary Incontinence in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Completes the Mind Over Matter; Healthy Bowels, Healthy Bladder workshop in the spring 2017.
  Interventions: Behavioral: Mind Over Matter; Healthy Bowels, Healthy Bladder
- Control (Other): Completes the Mind Over Matter; Healthy Bowels, Healthy Bladder workshop in the fall 2017.
  Interventions: Behavioral: Mind Over Matter; Healthy Bowels, Healthy Bladder

INTERVENTIONS:
Behavioral: Mind Over Matter; Healthy Bowels, Healthy Bladder — This three-session workshop is based on proven principles of behavior change addressing urinary and bowel continence self-management and health education and has been developed specifically for administration to women age 50 and older in senior centers.

SUMMARY:
The goal of this study is to obtain data about the effectiveness, reach, adoption, and implementation potential of an innovative, combined urinary/bowel continence workshop through a randomized controlled trial in six Wisconsin communities. This three-session workshop is based on proven principles of behavior change addressing urinary and bowel continence self-management and health education and has been developed specifically for administration to women age 50 and older in senior centers. We hypothesize that workshop participants will experience improvements in urinary and bowel incontinence symptoms, will have increased levels of care-seeking and self-efficacy for these conditions, and will maintain the self-management strategies taught in the workshop 3 months following completion of the workshop. We further hypothesize that this workshop will reach its intended target population (independent senior women with incontinence) and will improve their mental health by destigmatizing the condition of incontinence.

ELIGIBILITY:
Inclusion Criteria:

* qualifying symptoms within last 3 months
* able to speak English
* lives independently

Exclusion Criteria:

* new treatment for target symptoms within last 3 months

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 122 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Symptom Improvement | 3 months after treatment group completes intervention
  Patient Global Impression of Improvement (PGI-I) regarding bladder or bowel incontinence

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory-20 | 3 months after treatment group completes intervention
  validated instrument
Geriatric Self-Efficacy for Urinary Incontinence (GSE-UI) | 3 months after treatment group completes intervention
  validated instrument
Barriers to Care-seeking for Accidental Bowel Leakage (BCABL) | 3 months after treatment group completes intervention
  validated instrument
Barriers to Incontinence Care-seeking (BICS-Q) | 3 months after treatment group completes intervention
  validated instrument

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Brown, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown HW, Braun EJ, Wise ME, Myers S, Li Z, Sampene E, Jansen SM, Moberg DP, Mahoney JE, Rogers RG. Small-Group, Community-Member Intervention for Urinary and Bowel Incontinence: A Randomized Controlled Trial. Obstet Gynecol. 2019 Sep;134(3):600-610. doi: 10.1097/AOG.0000000000003422. PMID 31403596